CLINICAL TRIAL: NCT06363760
Title: A Long-Term Follow-Up Study of Participants With Sickle Cell Disease or Transfusion Dependent β-Thalassemia Who Received EDIT-301
Status: Enrolling by invitation | Type: Observational
Sponsor: Editas Medicine, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EDIT-301-LTFU-001
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Disease; Transfusion-dependent Beta-Thalassemia; Hemoglobinopathies
Keywords: Sickle Cell Disease; Sickle Cell Anemia; Sickling Disorder Due to Hemoglobin S; Beta-Thalassemia; Thalassemia Major; Thalassemia Intermedia; Hemoglobinopathies; CRISPR-Cas12a; Autologous CD34+; Genetic Diseases, Inborn; Hematologic Diseases; Anemia; Anemia, Hemolytic, Congenital; Anemia, Hemolytic
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinopathies; beta-Thalassemia; Genetic Diseases, Inborn; Hematologic Diseases; Anemia; Anemia, Hemolytic, Congenital; Anemia, Hemolytic | interventions — Safety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: All participants who complete or discontinue one of the parent studies (EM-SCD-301-001 or EDIT-301-BThal-001)
  Interventions: Other: Safety and efficacy assessments

INTERVENTIONS:
Other: Safety and efficacy assessments — Assessed throughout the duration of the study.

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of EDIT-301 in participants with severe sickle cell disease (SCD) or transfusion-dependent β-thalassemia (TDT) who have received EDIT-301.

DETAILED DESCRIPTION:
This is a non-interventional, multicenter study evaluating the long-term safety and efficacy of EDIT-301 in participants with severe sickle cell disease (SCD) or transfusion dependent b-thalassemia (TDT) who received EDIT-301 in parent studies EM-SCD-301-001 (NCT04853576) or EDIT-301-BThal-001 (NCT05444894). No investigational drug product will be administered in the LTFU study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have received an EDIT-301 infusion as part of a clinical study.
* Participant or legal representative/guardian (if applicable) must sign and date the informed consent form (ICF) or assent, if applicable for this long-term follow-up study.

Exclusion Criteria:

* Participant is still actively enrolled in an EDIT-301 treatment study and has not yet met eligibility for long term follow-up in this study.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will be subjects currently enrolled in any one of the two parent studies ( EM-SCD-301-001 or EM-301-BThal-001)
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2040-08 (Estimated); Study Completion 2040-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events of special interest (AESI) | up to 15 years post EDIT-301 infusion
Adverse events of interest (AEI) | up to 15 years post EDIT-301 infusion
All-cause mortality | up to 15 years post EDIT-301 infusion
Adverse events (AEs) related to EDIT-301 | up to 15 years post EDIT-301 infusion
Serious adverse events (SAEs) | up to 15 years post EDIT-301 infusion

SECONDARY OUTCOMES:
Proportion of SCD participants with severe vaso-occlusive events (sVOEs) over time post-EDIT-301 infusion | up to 15 years post EDIT-301 infusion
Proportion of SCD participants with vaso-occlusive events (VOEs) over time post-EDIT-301 infusion | up to 15 years post EDIT-301 infusion
Frequency of SCD-related transfusions over time post-EDIT-301 infusion for SCD participants | up to 15 years post EDIT-301 infusion
Proportion of TDT participants with sustained transfusion independence (TI) over time | up to 15 years post EDIT-301 infusion
Proportion of TDT participants with sustained transfusion reduction (TR) over time | up to 15 years post EDIT-301 infusion
Frequency of TDT-related transfusions over time post-EDIT-301 infusion for TDT participants | up to 15 years post EDIT-301 infusion
SCD and TDT: Percent of peripheral red blood cells (RBCs) containing HbF (F-cells) over time | up to 15 years post EDIT-301 infusion
SCD and TDT: Total hemoglobin (Hb) concentration (g/dL) over time | up to 15 years post EDIT-301 infusion
SCD and TDT: Proportion of alleles with intended genetic modification present in peripheral blood nucleated cells and bone marrow derived CD34+ over time | up to 15 years post EDIT-301 infusion
Average HbF (pg) per RBC over time for SCD participants | up to 15 years post EDIT-301 infusion
Complete Blood Count (CBC) red cell indices assay over time for SCD participants | up to 15 years post EDIT-301 infusion
Average HbF (pg) per F-cell over time for SCD participants | up to 15 years post EDIT-301 infusion
HbF and HbS concentration (g/dL) over time for SCD participants | up to 15 years post EDIT-301 infusion
The level of HbF production determined by fractionation of different forms of Hb (including but not limited to HbA, HbA2, HbC, HbD, HbE, and HbS) over time for SCD participants. | up to 15 years post EDIT-301 infusion
Percentage of HbF over total non-transfused total Hb (non-transfused total Hb refers to the total g/dL of all Hb variants, excluding HbA) over time for TDT participants. | up to 15 years post EDIT-301 infusion
HbF concentration (g/dL) over time for TDT participants | up to 15 years post EDIT-301 infusion
Iron overload of TDT participants | up to 15 years post EDIT-301 infusion
  As measured by a) Liver iron concentration (LIC) as assessed by R2* magnetic resonance imaging (MRI) for the first 3 years in this study; b) Cardiac iron concentration (CIC) as assessed by T2* MRI for the first 3 years of this study; c) Serum ferritin levels over time.
Proportion of TDT participants receiving iron chelation therapy over time. | up to 15 years post EDIT-301 infusion

CONTACTS AND LOCATIONS:
Locations (18):
- United States (16):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Smilow Cancer Hospital, New Haven, Connecticut
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University Medical Center - Department of Pediatrics, New York, New York
  - Columbia University Medical Center, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Tristar Medical Group Children's Specialists/Sarah Cannon Center for Blood Cancers, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Cook Children's, Fort Worth, Texas
- Canada (2):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Princess Margaret Cancer Centre-University Health Network, Toronto, Ontario